CLINICAL TRIAL: NCT00826241
Title: A Phase II Study of Dose-Dense Temozolomide and Lapatinib for Recurrent Low-Grade and Anaplastic Supratentorial, Infratentorial and Spinal Cord Ependymoma
Brief Title: Dose-Dense Temozolomide + Lapatinib for Recurrent Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: CERN Foundation - Collaborative Ependymoma Research Network (Network)
Responsible Party: Principal Investigator, Mark Gilbert, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 999916005; NCI-2012-02131 (Other: NCI); 16-C-N005 (Other: NIH)
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Brain Tumors; Spinal Cord Tumors
Keywords: Brain Tumor; Central Nervous System; CNS; Spinal Cord Tumor; Anaplastic Ependymoma; Supratentorial Ependymoma; Infratentorial Ependymoma; Spinal Cord Ependymoma; Lapatinib; GW572016; Temozolomide; Temodar
MeSH Terms: conditions — Brain Neoplasms; Spinal Cord Neoplasms; Ependymoma | interventions — Temozolomide; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temozolomide + Lapatinib (Experimental): Temozolomide starting dose 125 mg/m^2 daily by mouth on days 1-7 & 15-21 of a 28 day cycle. Lapatinib starting dose 1250 mg daily by mouth.
  Interventions: Drug: Temozolomide; Drug: Lapatinib

INTERVENTIONS:
Drug: Temozolomide — Starting dose 125 mg/m^2 daily by mouth on days 1-7 & 15-21 of a 28 day cycle.
  Other Names: Temodar
Drug: Lapatinib — Starting dose 1250 mg daily by mouth.
  Other Names: GW572016

SUMMARY:
The goal of this clinical research study is to learn if lapatinib when given in combination with temozolomide can help to control ependymoma that has come back after treatment. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Temozolomide is designed to kill cancer cells by damaging deoxyribonucleic acid (DNA) (the genetic material of cells). This could cause the tumor cells to die.

Lapatinib is designed to prevent or slow down the growth of cancer cells by blocking proteins inside the cancer cell, called the human epidermal growth factor receptor 2 (Her2/neu) receptor and the epidermal growth factor receptor (EGFR).

Study Drug Administration:

If you are found to be eligible to take part in this study, every day, you will take lapatinib by mouth once a day in the morning. You should take lapatinib 1 hour before or 1 hour after eating, with at least 1 cup (about 8 oz.) of water.

On Days 1-7 and 15-21 of each cycle, you will take temozolomide by mouth 1 time each day. You will start to take a lower dose of temozolomide for the first 2 cycles, then take a higher dose for Cycles 3 and beyond if you tolerate the treatment. It should be taken at least 2 hours before and 2 hours after eating with 1 cup (about 8 oz.) of water.

You should swallow temozolomide and/or lapatinib whole, one right after the other, without chewing either of the study drugs. If you vomit while taking temozolomide and lapatinib, you cannot take more capsules before the next scheduled dose. You should report any missed pills or trouble you have with taking the pills to your study doctor. Your study doctor will give you a form (patient diary) to fill out to keep track of your treatment. You will be asked to return your completed diary and pill bottles at each visit with your doctor.

Each study "cycle" is 28 days.

Study Visits:

Every 2 weeks, blood (about 2-3 teaspoons) will be drawn for routine tests and to check your blood's ability to clot.

Every 8 weeks, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a neurological exam.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will complete the quality of life questionnaire.
* You will have an magnetic resonance imaging (MRI) scan to check the status of the disease.
* You will have either a multi-gated acquisition scan (MUGA) scan (if the doctor thinks it is needed) or an echocardiogram.

Length of Study:

You will be on study treatment for up to 2 years. You will be taken off study treatment early if the disease gets worse or you experience intolerable side effects.

After you are off study, you may be able to continue taking lapatinib for as long as the doctor thinks it is in your best interest. Your doctor will discuss this with you.

End-of-Study Visit:

After you go off study treatment, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a neurological exam.
* Blood (about 3 teaspoons) will be drawn for routine tests and to check your blood's ability to clot.
* You will complete the questionnaire.
* You will have an MRI scan to check the status of the disease.
* You will have either a MUGA scan (if the doctor thinks it is needed) or an echocardiogram.

Long-Term Follow-up Visit:

If you go off treatment (having completed the maximum 24 months on study drug treatment) and have stable disease or response, you will have an MRI scan to check the status of the disease every 2 months for first year after you are off study, then every 3 months for the second year, then every 4 months for the third year, and then every 6 months from then on.

If you continue taking lapatinib after you have completed up to 24 months on study treatment, you will have a clinic visit and an MRI scan to check the status of the disease every 2 months for as long as the doctor thinks it is needed. At the clinic visits, you will be asked how you are doing.

If you went off study treatment because the disease got worse or you experienced intolerable side effects, after the end-of-study visit, the study staff will call you every 3 months from then on to check how you are doing. Each phone call will take about 5 minutes.

This is an investigational study. Temozolomide is Food and Drug Administration (FDA) approved or commercially available for the treatment of tumors of the nervous system. Lapatinib is FDA approved and commercially available for the treatment of breast cancer. However, lapatinib is not FDA approved for the treatment of brain tumors. The use of lapatinib with temozolomide in the treatment of brain tumors and spinal tumors is investigational.

Up to 50 patients will take part in this multicenter study. Up to 30 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven ependymoma or anaplastic ependymoma. There must be pathologic or imaging confirmation of tumor progression or regrowth. The patients histologic diagnosis must be confirmed on Central Pathology Review prior to registration Step 2.
2. History and physical examination, including neurologic examination, within 2 weeks prior to registration.
3. Patients must be able to undergo brain or spine magnetic resonance imaging (MRI) scans with intravenous gadolinium, based on tumor location(s) within 14 days prior to registration.
4. Patients must be on a steroid dose that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required.
5. Karnofsky performance status >/= 70
6. Age >/= 18
7. Complete blood count (CBC)/differential obtained within 14 days prior to registration, with adequate bone marrow function defined as follows: 1) Absolute neutrophil count (ANC) >/= 1,500/mm^3. 2) Platelets >/= 100,000 cells/mm^3. 3) Hemoglobin >/= 10.0 gm/dL (Note: The use of transfusion or other intervention to achieve Hgb >/= 10.0 is acceptable). 4) White blood cell count (WBC) >/= 3,000/mcL.
8. Adequate liver function within 14 days prior to registration, defined as follows: serum glutamic pyruvic transaminase (SGPT) [alanine aminotransferase (ALT)] < 2.5 times the upper limit of normal, Bilirubin </= 1.6 mg/dL
9. Adequate renal function within 14 days prior to registration, defined as follows: Creatinine < 1.7 mg/dL
10. Patients must have recovered from the toxic effects of prior therapy, and there must be a minimum time of: 1) 28 days from the administration of any investigational agent. 2) 28 days from administration of prior cytotoxic therapy with the following exceptions: (a) 14 days from administration of vincristine. (b) 42 days from administration of nitrosoureas. (c) 21 days from administration of procarbazine.
11. ( 11. continued) 3) 7 days from administration of non-cytotoxic agents [e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count)]. 4) 28 days from prior radiation therapy.
12. Patients must have recovered from the effects of surgery and a minimum of 14 days must have elapsed from the day of surgery to the day of registration. For core or needle biopsy, a minimum of 7 days must have elapsed prior to registration.
13. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, an MRI should be done no later than 96 hours in the immediate postoperative period or at least 4 weeks postoperatively, within 14 days prior to registration. If the " within 96-hour of surgery " scan is more than 14 days before registration, the scan needs to be repeated.
14. Patients must sign study-specific informed consent and authorization for the release of their protected health information prior to registration. Patients must be registered in the MD Anderson Cancer Center Office of Multicenter Clinical Research (MDACC OMCR) database prior to treatment with study drug.
15. Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 14 days prior to registration.
16. Women of childbearing potential and male participants must practice adequate contraception
17. All patients must have an left ventricular ejection fraction (LVEF) measurement of at least 50% by Echo or MUGA (if clinically indicated) within 14 days prior to registration. The method used for LVEF assessment in an individual subject must be the same throughout the trial.

Exclusion Criteria:

1. Prior invasive malignancy that is not the ependymoma (except non-melanomatous skin cancer or carcinoma in situ of the cervix) unless the patient has been disease free and off therapy for that disease for a minimum of 3 years
2. Transmural myocardial infarction or unstable angina within 3 months prior to study registration
3. Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >/= 2 mm using the analysis of an electrocardiography (EKG) performed within 14 days prior to registration
4. New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration
5. History of stroke or transient ischemic attack within 3 months prior to registration.
6. Inadequately controlled hypertension (systolic blood pressure > 140 mm Hg and/or diastolic blood pressure > 90 mm Hg despite antihypertensive medication)
7. History of cerebral vascular accident (CVA) within 3 months prior to registration
8. Serious and inadequately controlled cardiac arrhythmia
9. Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection)
10. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
11. Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with acquired immunodeficiency syndrome (AIDS) from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
12. Pregnant or nursing women because of concern of fetal/infant exposure to these agents
13. Any condition that impairs ability to swallow pills (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, active peptic ulcer disease).
14. Patients cannot be receiving enzyme-inducing anti-epileptic Drugs (EIAEDs) nor any other Image result for CYP3A4 Cytochrome P450 3A4 (CYP3A4) inducers such as rifampin or St. John's wort beginning at least 14 days prior to registration Step 2.
15. Patients cannot be receiving CYP3A4 inhibitors beginning at least 7 days prior to registration Step 2.
16. Patients must not have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
17. Patients cannot be receiving HAART (Highly Active Anti-Retroviral Therapy) therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Penas-Prado, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide + Lapatinib
Started | 58
Completed | 31
Not Completed | 27
Not completed — Withdrawal from Follow-up | 1
Not completed — Withdrew consent | 2
Not completed — Death | 4
Not completed — Non-reportable(not qualify as Gr. 5 SAE) | 1
Not completed — Non-compliance | 1
Not completed — Progression of disease | 1
Not completed — Patient refused follow-up | 3
Not completed — Lost to Follow-up | 9
Not completed — Could not obtain records | 1
Not completed — Screen failure | 2
Not completed — Pt unable to proceed to registration | 1
Not completed — Pt opt not to proceed w/trmt | 1

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide + Lapatinib
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.77 (15.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 58
  American Indian/Alaskan Native | 1
  Black | 2
  White | 51
  Unknown | 3
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression defined as progressive disease, toxicity at a level of severity that precludes the patient continuing on the protocol, or death. Progression is a 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Assessed every two months till disease progression, up to 4 years
Population: 8 patients were not evaluable/replaced: 2 - withdrew,1 - non-compliant, 2 - screen failures, 1 - could not obtain records, 1 - opted not to proceed with treatment, and 1 - unable to proceed to registration.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temozolomide + Lapatinib
Number analyzed (Participants) | 50
Months | 7.8 [5.2 to 12.2]

2. Secondary Outcome: Number of Participants With an Overall Response (Complete Response or Partial Response) Assessed by the MacDonald Criteria
Description: Anti-tumor activity as determined by the overall response (Complete response (CR) or partial response (PR)) was assessed by the MacDonald criteria. Complete response is complete resolution of all lesions. The patient cannot be on any corticosteroids with the exception of adrenal replacement doses. Partial response is ≥50% reduction in the sum of products of all measurable lesions over baseline sum observed using the same techniques as baseline. The patient must be on a stable or decreased dose of corticosteroids to be evaluable for response.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide + Lapatinib
Number analyzed (Participants) | 50
Participants
  Complete Response | 2
  Partial Response | 8

3. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 111 months and 26 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Temozolomide + Lapatinib
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 111 months and 26 days.
Description: 8 patients were not evaluable/replaced: 2 - withdrew,1 - non-compliant, 2 - screen failures, 1 - could not obtain records, 1 - opted not to proceed with treatment, and 1 - unable to proceed to registration.
Arm/Group | Temozolomide + Lapatinib
All-Cause Mortality (participants affected / at risk) | 4/50
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide + Lapatinib (N=50)
Ataxia (incoordination) (Nervous system disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hemorrhage, GU : Bladder (Gastrointestinal disorders) | 1 (2)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Surgical and medical procedures) | 1 (2)
Infection (Infections and infestations) | 2 (4) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) : Skin (cellulitis)
Infection with normal ANC or Grade 1 or 2 neutrophils : Skin (cellulitis) (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : Urinary tract NOS (Infections and infestations) | 1 (2)
Leukocytes (total WBC) (Investigations) | 1 (2)
Lymphopenia (Investigations) | 2 (18)
Muscle weakness, generalized or specific area (not due to neuropathy) : Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (2)
Pain - Other (Specify, left hip) (Musculoskeletal and connective tissue disorders) | 1 (2)
Platelets (Investigations) | 2 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (2)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (2) — upper respiratory congestion -stable bronchitis vs pneumonia
Secondary Malignancy - possibly related to cancer treatment (Specify,B-cell/large cell lymphoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide + Lapatinib (N=50)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (20)
Alkaline phosphatase (Investigations) | 7 (18)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Allergy/Immunology - Other (Specify, environmental allergic dry cough) (Immune system disorders) | 1 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 17 (54)
Amylase (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 10 (22)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 16 (50)
Ataxia (incoordination) (Nervous system disorders) | 6 (14)
Auditory/Ear - Other (Specify, fluttering sensation) (Ear and labyrinth disorders) | 1 (2)
Auditory/Ear - Other (Specify, hearing loss; present at baseline) (Ear and labyrinth disorders) | 1 (2)
Bicarbonate, serum-low (Investigations) | 1 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 4 (16)
Blood/Bone Marrow - Other (Specify, BUN) (Blood and lymphatic system disorders) | 1 (2)
Blood/Bone Marrow - Other (Specify,elevated bilirubin) (Blood and lymphatic system disorders) | 1 (2)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (20)
Cardiac General - Other (Specify, sinus tachycardia) (Cardiac disorders) | 1 (2)
Cataract (Eye disorders) | 1 (2)
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (2)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 3 (6)
Cognitive disturbance (Nervous system disorders) | 4 (8)
Confusion (Psychiatric disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 32 (82)
Constitutional Symptoms - Other (Specify, constipation) (General disorders) | 1 (2)
Constitutional Symptoms - Other (Specify, fatigue) (General disorders) | 1 (2)
Constitutional Symptoms - Other (Specify, hyposmia: reduced ability to smell) (General disorders) | 1 (2)
Constitutional Symptoms - Other (Specify,insomnia) (General disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (18)
Creatinine (Investigations) | 6 (22)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (4)
Dermatology/Skin - Other (Specify, _) (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin - Other (Specify,steroid-related acne) (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatology/Skin - Other (Specify, paresthesia) (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 19 (46) — Herpes Zoster - pain around bra line w/ out rash. Has Zoster before in same area.
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (4)
Dizziness (Nervous system disorders) | 5 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (6)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 (24)
Edema: head and neck (General disorders) | 2 (4)
Edema: limb (General disorders) | 8 (18)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (2)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 18 (42)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 39 (102)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (14)
Flatulence (Gastrointestinal disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (2)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (4)
Gastrointestinal - Other (Specify, abdominal distension) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal - Other (Specify, cramps in pelvis) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal - Other (Specify,gastrointestinal pain (intermittent)) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal - Other (Specify, mucositis oral) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal - Other (Specify, rectal discomfort) (Gastrointestinal disorders) | 1 (2)
Gastrointestinal - Other (Specify, stool incontinence) (Gastrointestinal disorders) | 1 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 22 (86)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 9 (24)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (8)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 2 (4)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 2 (4)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (4)
Hemoglobin (Investigations) | 25 (190)
Hemorrhage, GI : Lower GI NOS (Gastrointestinal disorders) | 1 (2)
Hemorrhage, GI : Oral cavity (Gastrointestinal disorders) | 1 (2)
Hemorrhage, GI : Rectum (Gastrointestinal disorders) | 2 (4)
Hemorrhage/Bleeding - Other (Specify, gums) (Gastrointestinal disorders) | 2 (4)
Hemorrhage/Bleeding - Other (Specify, nose) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Surgical and medical procedures) | 1 (2)
Hot flashes/flushes (Vascular disorders) | 2 (4)
Hypertension (Vascular disorders) | 4 (8)
Hypotension (Vascular disorders) | 1 (2)
Incontinence, anal (Gastrointestinal disorders) | 4 (8)
Incontinence, urinary (Renal and urinary disorders) | 6 (14)
Infection - Other (Specify, bronchial infection) (Infections and infestations) | 1 (2)
Infection - Other (Specify,Other, toe fungal) (Infections and infestations) | 1 (2)
Infection - Other (Specify,shingles) (Infections and infestations) | 3 (6)
Infection - Other (Specify, Varicella Zoster) (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : Esophagus (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : External ear (otitis externa) (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (2) — Foreign body (e.g., graft, implant, prosthesis, stent)
Infection with normal ANC or Grade 1 or 2 neutrophils : Skin (cellulitis) (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : Upper airway NOS (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : Urinary tract NOS (Infections and infestations) | 4 (10)
Infection with unknown ANC : Bladder (urinary) (Infections and infestations) | 1 (2)
Infection with unknown ANC : Urinary tract NOS (Infections and infestations) | 2 (4)
Insomnia (Psychiatric disorders) | 7 (14)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 30 (352)
Libido (Reproductive system and breast disorders) | 1 (2)
Lipase (Investigations) | 1 (2)
Lymphatics - Other (Specify, left thigh) (Blood and lymphatic system disorders) | 1 (2)
Lymphatics - Other (Specify,mild peripheral edema) (Blood and lymphatic system disorders) | 1 (2)
Lymphopenia (Investigations) | 35 (444)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (8)
Memory impairment (Nervous system disorders) | 11 (22)
Metabolic/Laboratory - Other (Specify, Akaline Phosphatase Serum Low) (Metabolism and nutrition disorders) | 2 (4)
Metabolic/Laboratory - Other (Specify, Albumin serum high) (Metabolism and nutrition disorders) | 5 (10)
Metabolic/Laboratory - Other (Specify,alkaline phosphatase count low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify,amylase serum low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify,AST-SGOT serum low) (Metabolism and nutrition disorders) | 3 (6)
Metabolic/Laboratory - Other (Specify, BUN) (Metabolism and nutrition disorders) | 1 (6)
Metabolic/Laboratory - Other (Specify, BUN count increased) (Metabolism and nutrition disorders) | 2 (6)
Metabolic/Laboratory - Other (Specify, BUN serum high) (Metabolism and nutrition disorders) | 3 (12)
Metabolic/Laboratory - Other (Specify, BUN serum low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, carbon dioxide) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, carbon dioxide count increased) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, carbon dioxide serum high) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, chloride count decreased) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, chloride serum high) (Metabolism and nutrition disorders) | 5 (12)
Metabolic/Laboratory - Other (Specify, chloride serum low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, CO2 count increased) (Metabolism and nutrition disorders) | 2 (4)
Metabolic/Laboratory - Other (Specify, CO2 high serum) (Metabolism and nutrition disorders) | 6 (18)
Metabolic/Laboratory - Other (Specify, creatinine count decreased) (Metabolism and nutrition disorders) | 3 (6)
Metabolic/Laboratory - Other (Specify, creatinine serum low) (Metabolism and nutrition disorders) | 7 (16)
Metabolic/Laboratory - Other (Specify, CSF Total Nucleated Cells Increased) (Metabolism and nutrition disorders) | 2 (4)
Metabolic/Laboratory - Other (Specify, hyperalbumin) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, hyperphosphatemia) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, LDH) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, LDH serum increased) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, LDH count decreased) (Metabolism and nutrition disorders) | 2 (4)
Metabolic/Laboratory - Other (Specify, LDH count increased) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, LDH serum high) (Metabolism and nutrition disorders) | 3 (8)
Metabolic/Laboratory - Other (Specify, LDH serum low) (Metabolism and nutrition disorders) | 2 (10)
Metabolic/Laboratory - Other (Specify, phosphorous serum high) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, protein count decreased) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, protein serum low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, SGOT decreased count) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, total protein serum low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, uric acid serum low) (Metabolism and nutrition disorders) | 1 (2)
Metabolic/Laboratory - Other (Specify, vitamin B12 deficiency) (Metabolism and nutrition disorders) | 1 (2)
Mood alteration : (Psychiatric disorders) | 1 (2)
Mood alteration : Agitation (Psychiatric disorders) | 2 (4)
Mood alteration : Anxiety (Psychiatric disorders) | 9 (18)
Mood alteration : Depression (Psychiatric disorders) | 6 (14)
Mucositis/stomatitis (clinical exam) : (Gastrointestinal disorders) | 1 (2)
Mucositis/stomatitis (clinical exam) : Oral cavity (Gastrointestinal disorders) | 1 (2)
Mucositis/stomatitis (functional/symptomatic) : Oral cavity (Gastrointestinal disorders) | 2 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) : Extremity-lower (Musculoskeletal and connective tissue disorders) | 7 (16)
Muscle weakness, generalized or specific area (not due to neuropathy) : Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) : Facial (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness, generalized or specific area (not due to neuropathy) : Left-sided (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) : Right-sided (Musculoskeletal and connective tissue disorders) | 5 (10)
Muscle weakness, generalized or specific area (not due to neuropathy) : Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3 (6)
Musculoskeletal/Soft Tissue - Other (Specify, difficulty walking) (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal/Soft Tissue - Other (Specify, intermittent back pain) (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal/Soft Tissue - Other (Specify, left hand) (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal/Soft Tissue - Other (Specify, lower extremity) (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal/Soft Tissue - Other (Specify, paresthesia, left hand (carpal tunnel type syndrome) (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal/Soft Tissue - Other (Specify, right back tightness) (Musculoskeletal and connective tissue disorders) | 1 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (4)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 32 (82)
Neurology - Other (Specify, __) (Nervous system disorders) | 12 (32)
Neuropathy: cranial : CN VII Motor-face; Sensory-taste (Nervous system disorders) | 2 (4)
Neuropathy: cranial : CN VIII Hearing and balance (Nervous system disorders) | 1 (2)
Neuropathy: motor (Nervous system disorders) | 6 (12)
Neuropathy: sensory (Nervous system disorders) | 22 (52)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 17 (154)
Obstruction, GU : Prostate (Reproductive system and breast disorders) | 1 (2)
Ocular/Visual - Other (Specify, Dysconjugate gaze. Present after surgery.) (Eye disorders) | 1 (2)
Ocular/Visual - Other (Specify, left hemaniopsia) (Eye disorders) | 1 (2)
Ocular/Visual - Other (Specify, vision loss left eye) (Eye disorders) | 1 (2)
Ocular/Visual - Other (Specify, visual impairment) (Eye disorders) | 1 (2)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 2 (4)
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1 (2)
Pain (General disorders) | 1 (2)
Pain - Other (Specify, back and right arm) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, headaches) (Nervous system disorders) | 1 (2)
Pain - Other (Specify, joint pain) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, left anterior iliac spine) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, left leg) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, left sacrum pain) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, leg pain) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, musculoskeletal-back) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, neuralgia) (Nervous system disorders) | 1 (2)
Pain - Other (Specify, pain in the rash area chest and the back) (Skin and subcutaneous tissue disorders) | 1 (2)
Pain - Other (Specify, pain-pelvis) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, RUQ) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, severe pain left thigh) (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Other (Specify, stomach pain) (Gastrointestinal disorders) | 1 (2)
Pain : Abdomen NOS (Gastrointestinal disorders) | 1 (2)
Pain : Back (Musculoskeletal and connective tissue disorders) | 13 (28)
Pain : Bone (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain : Breast (Reproductive system and breast disorders) | 1 (2)
Pain : Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 3 (6)
Pain : Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 (8)
Pain : Head/headache (Nervous system disorders) | 17 (38)
Pain : Joint (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain : Muscle (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain : Neck (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain : Oral cavity (Gastrointestinal disorders) | 1 (2)
Pain : Pain NOS (General disorders) | 1 (2)
Pain : Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain : Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Palpitations (Cardiac disorders) | 2 (4)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 (22)
Platelets (Investigations) | 23 (174)
Potassium, serum-high (hyperkalemia) (Investigations) | 3 (6)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (12)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 9 (22)
Pulmonary/Upper Respiratory - Other (Specify, sinus congestion) (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pyramidal tract dysfunction (Nervous system disorders) | 9 (18) — (e.g., increased tone, hyperreflexia, positive Babinski, decreased fine motor coordination)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 15 (48)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 16 (42)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 4 (8)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (4)
Renal/Genitourinary - Other (Specify, urinary tract infection) (Renal and urinary disorders) | 1 (4)
Rigors/chills (General disorders) | 2 (4)
Seizure (Nervous system disorders) | 3 (8)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (6)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 5 (10)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (18)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 5 (10)
Supraventricular and nodal arrhythmia : Atrial fibrillation (Cardiac disorders) | 1 (2)
Syncope (fainting) (Nervous system disorders) | 2 (4)
Syndromes - Other (Specify, tremors; left hand) (General disorders) | 1 (2)
Taste alteration (dysgeusia) (Eye disorders) | 1 (2)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (4)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 (2)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2 (4)
Tinnitus (Ear and labyrinth disorders) | 4 (8)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 (4)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 7 (26)
Urinary frequency/urgency (Renal and urinary disorders) | 7 (14)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 6 (12)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2)
Valvular heart disease (Cardiac disorders) | 1 (4)
Vision-blurred vision (Eye disorders) | 7 (14)
Vision-flashing lights/floaters (Eye disorders) | 1 (2)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 10 (24)
Weight loss (Investigations) | 9 (18)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT00826241/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT00826241/ICF_001.pdf